CLINICAL TRIAL: NCT02065193
Title: Social Communication Research and Epidemiological Study in China
Brief Title: Prevalence of Autism Spectrum Conditions in Mainland China
Acronym: China SCORE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Cambridge (Other)
Collaborators: China Disabled Persons Federation (Other Government); Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Sophia Xiang Sun, Cambridge-CUHK International Fellow, Chinese University of Hong Kong
Other Study IDs: China SCORE study
Record Dates: First submitted 2014-02-12; First posted 2014-02-17 (Estimated); Last update posted 2014-02-17 (Estimated); Status verified 2014-02

CONDITIONS: Autism Spectrum Conditions/Disorders
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (14):
- Beijing group
  Interventions: Behavioral: ADOS/ADI-R/Clinical assessment
- Guangdong group
  Interventions: Behavioral: ADOS/ADI-R/Clinical assessment
- Shenzhen group
  Interventions: Behavioral: ADOS/ADI-R/Clinical assessment
- Shanxi group
  Interventions: Behavioral: ADOS/ADI-R/Clinical assessment
- Liaoning group
  Interventions: Behavioral: ADOS/ADI-R/Clinical assessment
- Jilin group
  Interventions: Behavioral: ADOS/ADI-R/Clinical assessment
- Heilongjiang group
  Interventions: Behavioral: ADOS/ADI-R/Clinical assessment
- Jiangsu group
  Interventions: Behavioral: ADOS/ADI-R/Clinical assessment
- Zhejiang group
  Interventions: Behavioral: ADOS/ADI-R/Clinical assessment
- Fujian group
  Interventions: Behavioral: ADOS/ADI-R/Clinical assessment
- Henan group
  Interventions: Behavioral: ADOS/ADI-R/Clinical assessment
- Hubei group
  Interventions: Behavioral: ADOS/ADI-R/Clinical assessment
- Hunan group
  Interventions: Behavioral: ADOS/ADI-R/Clinical assessment
- 'Shanxi group
  Interventions: Behavioral: ADOS/ADI-R/Clinical assessment

INTERVENTIONS:
Behavioral: ADOS/ADI-R/Clinical assessment

SUMMARY:
The China SCORE study is a prevalence study of Autism Spectrum Conditions (ASC) in 14 regions in mainland China. It will include the following steps:

1. Large population-based screening This study will be conducted in urban areas but not rural areas across mainland China. One city of each region will participate, and in total there will be 14 cities for screening. Within each city, a number of 40 to 60 ordinary primary schools will be randomly selected from the defined region. All the students who are in 1st to 4th grade will asked to participate in order to form a sample of approximately 20,000 students.

   Screening questionnaires The screening pack includes the Chinese CAST, the AQ-Child, the AQ-Adult short version (10 items), and risk factors questionnaire. An information sheet and consent form will be included in the pack as well.
2. Further assessments We expect approximately 5% on the CAST will score positive in ordinary school population. Thus, for a 20,000 sample, we would expect 900 positives (90% response rate). All the screen-positives and a random selected 5% from borderline group will be invited for clinical assessment. The diagnosis of clinical assessment will be divided into three categories: definite ASC, suspected ASC, and non-ASC. Then all the children with clinical assessment results as definite ASC and suspected ASC and a randomly selected 10-20 non-ASC will be invited for research diagnostic assessment using the ADOS and ADI-R, as well as RPM as IQ test. After that, the consensus diagnosis between ADOS/ADI-R assessment and the clinical diagnosis will be the final diagnosis.
3. Case identification in special schools All the children in special schools or training institutes in study region will be asked to fill in the screening pack. The children who do not attend any ordinary or special schools will be identified according to their residential ID in the studied regions. All screen-positives in special education will be assessed using the ADOS and ADI-R. Then those who met the criteria of ASC on ADOS or/and ADI-R will be assessed by psychiatrists and the clinical diagnosis will be the final diagnosis.

If we combine the prevalence of ordinary schools and special schools together, we will get an estimate of the prevalence of ASC in school-population in China. If we combine all the cases identified from schools and from residential records, we will generate an estimate of the prevalence of ASC in the general population in mainland China.

ELIGIBILITY:
Inclusion Criteria:

* All children who are in study region will be recruited for this study.
* All children aged 6-11 years old.

Exclusion Criteria:

* Children who are not in the study region.
* Children who are not found from ordinary schools, private training centres, public special schools and community household with the help of local residence records will not be included for this study.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Study population in each city is a defined region, usually a district or two districts. We focus on urban populations in this study.
Sampling Method: Probability Sample
Enrollment: 280000 (Estimated)
Dates: Start 2013-04; Primary Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Three-staged consensus diagnosis | The assessments will be finished in one year.
  The prevalence of Autism Spectrum Conditions will be measured using screening and diagnostic instruments including the Childhood Autism Spectrum Test , the Autism Diagnostic Observation Schedule, the Autism Diagnostic Interview-Revised, and Clinical diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Carol Brayne, MD, Principal Investigator — University of Cambridge; Simon Baron-Cohen, PhD, Principal Investigator — University of Cambridge; Carrie Allison, PhD, Principal Investigator — University of Cambridge; Hong You, MD, Principal Investigator — China Disabled Persons Federation; Jibin Han, Master, Principal Investigator — China Disabled Persons Federation; Sian Griffiths, MD, Principal Investigator — Chinese University of Hong Kong; Huso Yi, PhD, Principal Investigator — Chinese University of Hong Kong; Xiang Sun, PhD, Principal Investigator — Cambridge/CUHK; Fiona E Matthews, PhD, Principal Investigator — MRC Biostatistics Unit; Bonnie Auyeung, PhD, Principal Investigator — University of Cambridge
Locations (14):
- China (14):
  - Fujian CDPF, Fuzhou, Fujian
  - Shenzhen CDPF, Shenzhen, Guangdong
  - Heilongjiang CDPF, Jiamusi, Heilongjiang
  - Luoyang CDPF, Luoyang, Henan
  - Hengyang CDPF, Hengyang, Hunan
  - Jilin Mingzhi Centre, Jilin, Jilin
  - Liaoning CDPF, Benxi, Liaoning
  - Shanxi CDPF, Changzhi, Shanxi
  - Shanxi CDPF, Xian, Shanxi
  - Beijing CDPF, Beijing
  - Guangdong CDPF, Guangzhou
  - Zhejiang CDPF, Hangzhou
  - Hubei CDPF, Wuhan
  - Jiangsu CDPF, Yangzhou